CLINICAL TRIAL: NCT04327154
Title: A Prospective, Multicenter, Single-arm Clinical Trial Evaluating Safety and Performance of TISSIUMTM Nerve Coaptation Device for the Repair of Digital Nerve Discontinuities Where Gap Closure Can be Achieved by Flexion of the Extremity.
Brief Title: TISSIUM's Nerve Coaptation Device First-in-Human Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tissium (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PF00004-DC-2002
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-09

CONDITIONS: Digital Nerve Injury
Keywords: nerve repair; digital nerve repair; digital nerve lesion; peripheral nerve injury; peripheral nerve lesion; peripheral nerve repair
MeSH Terms: conditions — Peripheral Nerve Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital nerve repair (Experimental): There is no comparator for this study. All patients are in the treatment allocated group for digital nerve repair with the TISSIUM™ Nerve Coaptation Device.
  Interventions: Device: TISSIUM™ Nerve Coaptation Device

INTERVENTIONS:
Device: TISSIUM™ Nerve Coaptation Device — Placement of the TISSIUM™ Nerve Coaptation Device on repair site to achieve an end-to-end nerve coaptation.

SUMMARY:
The purpose of this study is to collect initial safety and device performance data of the TISSIUM's nerve coaptation device for the sutureless repair of digital nerve injuries of the hand in which there has been no substantial loss of nerve tissue. Additional clinical measures that assess device performance, use, and patient reported outcomes will be collected to guide future study design and potential device modifications.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing a repair of a proper digital nerve of the hand;
* 100% transection injury to the nerve under repair;
* Gap closure between the nerve ends can be achieved by flexion of the extremity without excessive tension;
* Clean surgical wound with sufficient healthy soft tissue that enables primary closure without adjunctive soft tissue procedures;
* Patient willing and able to provide a signed Patient Informed Consent Form;
* Patient willing and able to follow the study instructions and likely to complete all required study procedures and visits.

Exclusion Criteria:

* Patient has a known allergy to the constituent polymer of the investigational device;
* Patient has a documented diagnosis of peripheral neuropathy;
* Patient has a history of neuropathic pain;
* Patient has a history of injury to the nerve being studied;
* Patient has is missing the contralateral digit or with a history of injury to the contralateral digit (comparison control area);
* Patient is pregnant or nursing
* Any patient with a diagnosis of type 1 Diabetes Mellitus;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-12-16 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of complications (CIC) related to the investigational device | through 12-months post-procedure
  CIC includes the occurrence of any of the following complications:
  * Infection
  * Chronic pain (defined as pain lasting more than 3 months) not otherwise specified
  * Excessive inflammation as determined by the investigator
  * Device extrusion
  * Symptomatic neuroma formation
  * Impaired wound healing (examples are dehiscence, pain, skin irritation, keloid, scar hypertrophy)
  * Allergic reaction to the constituent polymer of the investigational device
  * Serious Adverse Device Effect (SADEs)

SECONDARY OUTCOMES:
Semmes-Weinstein monofilament (SWMF) for nerve functional recovery | at 6 months post-procedure
  Product performance will be assessed as functional nerve repair based on nerve functional recovery using Semmes-Weinstein monofilament (SWMF) at 6-months post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Randipsingh Bindra, Principal Investigator — Gold Coast University Hospital
Locations (2):
- Australia (2):
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Gold Coast University Hospital, Gold Coast, Queensland